CLINICAL TRIAL: NCT04550637
Title: A Multi-center Observative Study of Apixaban After Left Atrial Appendage Occlusion in Patients With Non-valvular Atrial Fibrillation
Brief Title: A Multi-center Study of Apixaban(APPROACH)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YL-2020-18
Record Dates: First submitted 2020-05-17; First posted 2020-09-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Evaluate the Safety and Efficacy of Apixaban
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anticoagulant therapy after percutaneous left atrial appendage: Oral apixaban
  Interventions: Drug: Oral apixaban

INTERVENTIONS:
Drug: Oral apixaban — apixaban (5 mg bid) is given until 12 weeks after surgery

SUMMARY:
The aim of the study is to enroll approximately 200 cases from 10 research centers nationwide, completed left atrial appendage occlusion (LAAO) successfully, and give apixaban (5 mg bid) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 85 years;
* understand the purpose of the trial, sign the informed consent form voluntarily
* successful surgery (no pericardial effusion, pericardial tamponade, or device displacement during operation; no pericardial effusion before discharge), meet COST standard during operation.
* In accordance with the indications for left atrial appendage occlusion: CHA2DS2-VAS2 score≥2 points and/or HAS-BLED score≥3 points
* unable or unwilling to take oral anticoagulants
* life expectancy≥1 year

Exclusion Criteria:

* History of previous cardiac surgery (valve disease, cardiomyopathy, severe coronary occlusion);
* Inability to tolerate trans-esophageal echocardiography;
* Preoperative trans-esophageal echocardiography suggests thrombus in left atrial appendage/left atrial;
* Patients with severe renal insufficiency (creatinine clearance rate<15ml/min);
* Patients with liver disease accompanied by abnormal blood coagulation and clinically related bleeding risks;
* Clinically significant active bleeding;
* The baseline platelet count is severely reduced: PLT≤50*10^9/L;
* Severe cardiac insufficiency (preoperative transthoracic echocardiography indicated LVEF <35%; uncontrolled heart failure (NYHA IV))
* Allergy or contraindication to anticoagulant drugs such as aspirin, clopidogrel, apixaban, etc .;
* Serious heart valve disease or other structural abnormalities need do elective surgical treatment; or severe coronary heart disease require limited-term intervention;
* Less than 45kg or more than 100kg.
* Take strong CYP3A4 and P-gp inhibitors (including pyrrole antifungal drugs, HIV protease inhibitors, etc.) for systemic treatment;
* Patients with other diseases besides atrial fibrillation (such as after mechanical valve replacement, spontaneous or recurrent venous thromboembolism, etc.) need anticoagulation treatment;
* Unsuccessful surgery (serious pericardial tamponade, massive bleeding and other life-threatening complications occur within 3 days after left atrial appendage closure);
* Pregnancy or lactation;
* Participating in other uncompleted clinical trials;
* Investigator considers inappropriate subjects.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is going to enroll approximately 200 cases who completed left atrial appendage occlusion (LAAO) successfully from 10 research centers nationwide.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse cardiovascular events | within 24 weeks after surgery
  all cause death, stroke, transient ischemic attack, systemic embolism

SECONDARY OUTCOMES:
Hemorrhagic/ischemic stroke events | within 24 weeks after surgery
  Stroke was defined as patients who developed dysarthria, aphasia, or weakness or sensory loss in the contralateral face, arm, or leg and cerebral ischemia and/or infarction. Diagnosis by clinical symptoms and cranial imaging examination.
Bleeding event | within 24 weeks after surgery
  Including dermal, mucosal, nasal, oral, gastrointestinal bleeding
Incidence of deaths | witnin 24 weeks after surgery
  All cause deaths (cardiac death, and non cardiac death)
Device related thrombosis | 12 weeks and 24 weeks after surgery
  Doctors find thrombosis after LAAC by transesophageal echocardiography.
Incidence of cardiovascular disease-related rehospitalization | 12 weeks and 24 weeks after surgery
  Cardiovascular disease include pericardial effusion, pericardial tamponade, poor cardiac function
severe adverse events | 12 weeks and 24 weeks after surgery
  Severe adverse events include re-inpatient for poor cardiac function and other severe adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, China